CLINICAL TRIAL: NCT00825656
Title: SINOL + MucoAd™ (SMAN) Evaluation Trial: A Double-Blind, Cross-Over Comparison of SINOL and SMAN in Subjects With Congestion Due to Allergic Rhinitis
Brief Title: Comparative Study of Sinol and Sinol-M in Patients With Congestion Due to Allergic Rhinitis
Acronym: SMAN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Strategic Biosciences (Industry)
Responsible Party: Martha WhiteMD, CPI, Institute for Asthma and Allergy
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMAN-0708
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Capsaicin; Homeopathic; Sinol; Sinol-M
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Sinol-M
  Interventions: Drug: Sinol or Sinol-M nasal spray
- 2 (Active Comparator): Sinol
  Interventions: Drug: Sinol or Sinol-M nasal spray

INTERVENTIONS:
Drug: Sinol or Sinol-M nasal spray — One spray in each nostril up to a maximum of 12 times / day on an "as needed" basis
  Other Names: Capsaicin nasal spray

SUMMARY:
The purpose of this study is to demonstrate the equivalence of two homeopathic capsaicin containing nasal sprays (Sinol-M™ and Sinol) in patients with nasal congestion due to allergic rhinitis.

DETAILED DESCRIPTION:
Sinol is an FDA registered, capsaicin-based, over-the-counter homeopathic nasal spray used for the relief of allergy and sinus conditions. It is an all-natural product that the patient uses on an as-needed basis for up to 12 times daily.

Sinol has been available in the US since 2004. In 2009 a second generation product, Sinol-M will be launched. Sinol-M is identical to the original formula but also contains MucoAd MucoAd™ is a patented non-toxic, non-irritating, liquid polymer mucoadhesive carrier that prolongs the contact time between drug and mucosa, thus increasing bioavailability. It can be loaded with nearly any pharmaceutical preparation and delivered a variety of mucosal tissues. Reduced mucociliary clearance of intranasally-applied drugs is desirable to reduce the naturally-occurring washing out of topically applied medications.

The objective of the current Phase IV, randomized, double-blind, cross-over study, was to evaluate the frequency of use and efficacy of SINOL and SINOL + MucoAd™ (Sinol-M) and to demonstrate non-inferiority of Sinol-M versus the existing product Sinol.

Additionally, as most homeopathic drugs are not supported by prospective clinical data there is a belief among many mainstream healthcare practitioners, and some consumers that these products do not work. This study therefore provides an opportunity to demonstrate improved efficacy versus no treatment (during the run-in and washout phases).

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate as indicated by providing written informed consent
* 12 years of age or older, of any gender and any race
* Have had a positive skin prick and/or intradermal test for a currently prevalent allergen within the past 5 years
* A history of allergic rhinitis, for at least 2 years
* Have undergone washout of all medications that could have an influence on the study
* Willing and able to make required study visits
* Able to follow instructions and record diary symptoms.
* Free of significant anatomic abnormalities, infection, bleeding, and mucosal ulcerations on nasal examination
* Have a TNSS between 4 and 12 averaged over the 7 days immediately prior to V2
* Have an average individual score for nasal congestion greater than or equal to 2 over the 7 days immediately prior to V2.

Exclusion Criteria:

* any concurrent disease that could interfere with the investigation or evaluation of the study medications such as: rhinitis medicamentosa or large obstructive nasal polyps
* any other anatomic nasal deformity that could interfere with their participation in the study
* asthma, with the exception of mild intermittent asthma
* congestion that, in the opinion of the study investigator, could interfere with successful nasal drug administration/absorption (in either nostril)
* use of systemic corticosteroids (oral, parenteral, intravenous, rectal) or inhaled or ocular corticosteroids within the last 30 days
* be undergoing allergy immunotherapy, unless on a stable dosing regimen throughout the course of the study
* Be using dermal potent or super-potent topical corticosteroids
* any systemic disorder that could interfere with the evaluation of the study medication
* hypersensitivity to the study drugs or any component thereof
* history of drug or alcohol abuse that would interfere with participation in the study
* history of severe, unstable, or uncontrolled cardiovascular, hepatic, renal and/or other diseases/illnesses that could be expected to interfere with the study
* upper or lower respiratory infection within 14 days of Vist 2
* acute sinusitis within 30 days of Visit 2
* any history or evidence of nasolacrimal drainage system malfunction
* Be planning to travel to an area significantly antigenically different for a substantial portion (more than 48 hours) of any given study week.
* participation in any other investigational study within 30 days before entry into this study or concomitantly with this study
* chronic or intermittent use of any prescription or over-the-counter (OTC) nasal spray during the study period

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Daily Total Nasal Symptom Score (congestion, rhinorrhea, sneezing, nasal itching) | twice daily for 28 days

SECONDARY OUTCOMES:
Number of sprays of study drug used | twice daily for 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Martha White, MD, Principal Investigator — Institute for Allergy and Asthma
Locations (1):
- Institute for Allergy and Asthma, Wheaton, Maryland, United States